CLINICAL TRIAL: NCT03616925
Title: Evaluation of Platelet Rich Fibrin Matrix(PRFM) as a Regenerative Material in Surgical Management of Human Periodontal Intraosseous Defects:A Randomized Controlled Trial
Brief Title: Evaluation of Platelet Rich Fibrin Matrix as Regenerative Material in Intraosseous Defects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: KLE Society's Institute of Dental Sciences (Other)
Responsible Party: Principal Investigator, Dr Laveena Singhal, Principal investigator, KLE Society's Institute of Dental Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KLESociety
Record Dates: First submitted 2018-04-08; First posted 2018-08-06 (Actual); Last update posted 2018-08-06 (Actual); Status verified 2018-08

CONDITIONS: Regenerative Inflammation

STUDY DESIGN:
Intervention Model Description: The patients for this study were selected from the outpatient section of the Department of Periodontics, KLE Society's institute of Dental Sciences, Bangalore, Karnataka. Fifteen patients, aged between 30-55 years (10 males and 5 females) diagnosed with chronic periodontitis, contributing to 30 sites were enrolled for the study by convenience sampling method. It was made clear to the potential subjects that participation was voluntary. Written informed consent was obtained from patients, and ethical clearance for the study was received from the Institutional Ethics Committee (IEC), KLE Society's institute of Dental Sciences, Bangalore. This Randomized controlled trial was carried out from November 2013 to October 2014.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Platelet rich fibrin matrix (Experimental): surgical open flap debridement with Application of Platelet rich fibrin matrix using Platelet Rich Fibrin Matrix kit in 15 intrabony defect sites
  Interventions: Biological: Platelet Rich Fibrin Matrix kit
- surgical open flap debridement (Active Comparator): only surgical open flap debridement was done without application of Platelet rich fibrin matrix in 15 intrabony defect sites
  Interventions: Procedure: surgical open flap debridement

INTERVENTIONS:
Biological: Platelet Rich Fibrin Matrix kit — Platelet Rich Fibrin Matrix kit was used to procure platelet rich fibrin matrix using centrifugation machine
  Other Names: centrifugation machine
  Arms: Platelet rich fibrin matrix
Procedure: surgical open flap debridement — only surgical open flap debridement was done without use of Platelet Rich Fibrin Matrix kit
  Arms: surgical open flap debridement

SUMMARY:
Technological advancement has led to the development of concentrated platelets, by means of centrifugation, popularly known as Platelet concentrates which seem to be a convenient approach to obtain autologous growth factors. Locally delivered platelet concentrates are supposed to increase the proliferation of connective tissue progenitors to stimulate fibroblast and osteoblast activity and enhance angiogenesis, all of which are fundamental to tissue healing and regeneration. Several techniques for platelet concentrates are available, each method leading to a different product with different biology and potential use. Different platelet concentrates are classified, depending on their leucocyte and fibrin content. Conventional platelet rich plasma (PRP), also known as first generation platelet concentrate is plasma with a platelet concentration above the normal physiologic levels found in blood.

Platelet Rich Fibrin Matrix (PRFM) is an autologous biologic material created by two step centrifugation of whole blood without the use of exogenous thrombin. Platelets isolated, remain intact and retain their growth factor compliment. This allows a more effective, sustained release of growth factors to the wound site following PRFM application. PRFM possesses the ability to enhance tissue repair by isolation, concentration and preservation of autologous platelets in a dense scaffold like fibrin matrix. The viable platelets contain intrinsic growth factors which are probably released in a desired spatial and temporal manner that affect every aspect of soft tissue and osseous healing.

Very limited studies have been conducted to assess the regenerative potential of this new modality i.e. PRFM. This study therefore aims at the evaluation of platelet rich fibrin matrix as a potential regenerative material in comparison with open flap debridement in human periodontal intraosseous defects.

DETAILED DESCRIPTION:
Periodontitis is a chronic inflammatory disease caused by bacterial Plaque, the onset and progression of which is modulated by a variety of risk factors such as systemic conditions and smoking. It causes pathological alterations of the periodontium, resulting in loss of connective tissue attachment to the tooth, apical migration of the junctional epithelium along the root surface and loss of supporting alveolar bone. If left untreated, cases of periodontal disease can lead to premature tooth loss. However, the complex structure of periodontium, which consist of soft connective tissue of gingiva and periodontal ligament, as well as the mineralized tissues, cementum and bone, makes periodontal wound healing a unique process.

Although, all the tissues of the periodontium get affected, the crux of the problem of chronic periodontal diseases lies in the changes that occur in the bone resulting in intraosseous defects of various architecture, the persistence of which even after completion of active periodontal treatment may increase the site-specific risk of progression of periodontitis.

The two primary components of periodontal therapy involves, the elimination of the periodontal infection by eliminating the pathogenic periodontal microflora which induces favourable clinical changes in the periodontium and substantial efforts should be made to alter the anatomic defect resulting from active periodontitis.

The resective surgical approach and mucogingival surgeries (MGS) were the major periodontal therapies until the 1970s. However, problems with esthetics, root sensitivity and root caries resulting from resective therapy for severe periodontitis were eventually pointed out. Also resective procedure was admitted to be a "Repair" and not "Regeneration" which has long been the goal of periodontal therapy. The past two decades has seen a radical change in periodontal surgery with a shift from resective periodontal surgery to regenerative therapies. Also the concept of treatment has changed towards regeneration with a goal of regaining natural periodontal apparatus.

Conventional surgical approaches (e.g., flap debridement) continue to offer time-tested and reliable methods to access root surfaces, reduce periodontal pockets and attain improved periodontal form/architecture. However, these techniques offer only limited potential to recover tissues, destroyed during earlier disease phases.

Broad ranges of treatment options are available, but only some are regarded as truly regenerative procedures. Periodontal regeneration is a complex process which requires an orchestrated sequence of biologic events, such as cell migration, adherence, growth, and differentiation involving a large number of growth factors and cytokines for its regulation.To accelerate clinical translation of the same, there is an ongoing need to develop therapeutics based on endogenous regenerative technology (ERT), which can stimulate latent self-repair mechanisms in patients and harness the host's innate capacity for regeneration. ERT in periodontics applies the patient's own regenerative 'tools', that is, patient-derived growth factors (GFs) and fibrin scaffolds, to create a material niche in an injured site where the progenitor/stem cells from neighbouring tissues can be recruited for (in situ) periodontal regeneration.

Growth factors are naturally occurring proteins that function in the body to promote the mitogenesis (proliferation), directed migration and metabolic activity of cells. Numerous growth factors have been identified, the expression of which following bone and soft tissue injury may regulate the repair and regenerative process. Platelets apart from their role in haemostasis have been reported to possess regenerative potential as their alpha granules are rich sources of various vital growth factors. These growth factors such as platelet derived growth factor, transforming growth factor β1, epithelial growth factor, vascular endothelial growth factor, insulin like growth factor and fibroblast growth factor whether used alone or in combination have been extensively studied and shown to promote the regeneration of oral and maxillofacial bone defects. Platelet growth factors may initiate healing by attracting undifferentiated cells within the fibrin matrix that is formed in the very early stages of healing process and by triggering cell division.

Technological advancement has led to the development of concentrated platelets, by means of centrifugation, popularly known as Platelet concentrates which seem to be a convenient approach to obtain autologous growth factors. Locally delivered platelet concentrates are supposed to increase the proliferation of connective tissue progenitors to stimulate fibroblast and osteoblast activity and enhance angiogenesis, all of which are fundamental to tissue healing and regeneration. Several techniques for platelet concentrates are available, each method leading to a different product with different biology and potential use. Different platelet concentrates are classified, depending on their leucocyte and fibrin content. Conventional platelet rich plasma (PRP), also known as first generation platelet concentrate is plasma with a platelet concentration above the normal physiologic levels found in blood.

Currently several methods are available for PRP preparation, most producing a liquid end product to promote tissue repair. Due to poor mechanical properties, conventional PRP is often difficult to handle in clinical settings that require secure implantation in a specific site or where released growth factors could be washed out during an operation. The physical properties of PRP can be changed if plasma and platelets are stimulated by the addition of calcium chloride and thrombin. The exogenous activation of platelets using bovine thrombin at the time of PRP preparation result in an almost immediate degranulation and disintegration of platelet granules. Consequently, complete growth factor release will take place at the time of PRP preparation and placement. Since wound healing requires a sequential appearance of vessels and cells over time, the immediate and almost complete release of platelet granules may have very little beneficial effect on later stages of healing.

In contrast, Platelet Rich Fibrin Matrix (PRFM) is an autologous biologic material created by two step centrifugation of whole blood without the use of exogenous thrombin. Platelets isolated, remain intact and retain their growth factor compliment. This allows a more effective, sustained release of growth factors to the wound site following PRFM application. PRFM possesses the ability to enhance tissue repair by isolation, concentration and preservation of autologous platelets in a dense scaffold like fibrin matrix. The viable platelets contain intrinsic growth factors which are probably released in a desired spatial and temporal manner that affect every aspect of soft tissue and osseous healing.

Very limited studies have been conducted to assess the regenerative potential of this new modality i.e. PRFM. This study therefore aims at the evaluation of platelet rich fibrin matrix as a potential regenerative material in comparison with open flap debridement in human periodontal intraosseous defects.

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy patients diagnosed with chronic periodontitis.
* Patients with bilateral infra bony pocket measuring ≥ 6mm with radiographic evidence of intrabony defect.

Exclusion Criteria:

* Pregnant /lactating women
* Patients taking any drug known to affect the number and function of platelets in the past 3 months.
* Patients with abnormal platelet count.
* Patients with immunologic diseases
* Current smokers.

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2014-09 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
the clinical change in regenerative potential of platelet rich fibrin matrix (PRFM) and open flap debridement (OFD) and OFD alone in periodontal defects. | baseline,3 months and 6 months
  Clinical parameters(plaque index, gingival index, probing pocket depth,attachment level)were combined to assess the change in the regenerative potential
Early wound healing index (EHI) was used to assess the wound healing potential of PRFM | 1 week
  Early wound healing index (EHI) was used to assess the wound healing potential of PRFM at 1 week.
change in the radiographic parameters in both the groups i.e,PRFM+OFD and OFD alone | baseline,3 months,6 months
  radiographic evidence of bilateral vertical osseous defects were categorized into test group [OFD + PRFM and control group [open flap debridement (OFD)]

CONTACTS AND LOCATIONS:
Overall Officials: Komal D Walia, MDS, Principal Investigator — KLE Society's Institute of Dental Sciences
Locations (1):
- Kle Society'S Institute of Dental Sciences, Bengaluru, Karnataka, India

IPD SHARING:
Plan to Share IPD: Undecided
except the results